CLINICAL TRIAL: NCT05763953
Title: The NODE-202 Study Multi-Center, Multi-National, Open-Label, Efficacy and Safety Study of Etripamil Nasal Spray in Pediatric Patients With Paroxysmal Supraventricular Tachycardia
Brief Title: The NODE-202 Study (Study of Etripamil Nasal Spray in Pediatric Patients)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Milestone Pharmaceuticals Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSP-2017-1265
Record Dates: First submitted 2023-02-03; First posted 2023-03-10 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Paroxysmal Supraventricular Tachycardia
Keywords: PSVT
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Etripamil NS 70mg (Experimental): Patients will be administered by study site personnel
  Interventions: Drug: Etripamil NS

INTERVENTIONS:
Drug: Etripamil NS — Part 1A: At least 12 patients will be administered with Etripamil NS (35 mg/100 μL per nostril) at a dose of 70 mg.
  Part 1B: At least 18 following patients will be administered with Etripamil NS at a dose determined by analysis of data generated from Part 1A.
  Part 2A: At least 12 patients will be administered with Etripamil NS at a dose selected based on appropriate body size-based modeling using PK assessments, as well as safety/tolerability, and efficacy data collected in Part 1.
  Part 2B: At least 18 following patients will be administered with Etripamil NS at a dose determined by analysis of data generated from Part 2A.

SUMMARY:
NODE-202 is a Phase 2, multicenter, multinational, single dose, open-label, 2-part, sequential design study in pediatric patients with an established diagnosis of paroxysmal supraventricular tachycardia (PSVT) presenting with a symptomatic episode of PSVT.

In Part 1, at least 30 patients aged 12 to <18 years will be enrolled and treated with etripamil nasal spray (NS). Efficacy, safety, tolerability and PK (for at least 12 patients) will be assessed after administration of 70 mg etripamil NS (Part 1A). At least 18 subsequent patients will be enrolled and treated with the etripamil NS with the dose determined by the Pharmacokinetic (PK) analysis and will undergo efficacy and safety/tolerability assessments (Part 1B).

In Part 2, at least 30 patients aged 6 to <12 years will be enrolled and treated with etripamil NS at a dose selected based on appropriate body size-based modeling, as well as efficacy, safety/tolerability, and PK data collected in Part 1. Efficacy, safety, tolerability and PK (for at least 12 patients) will be assessed after administration of etripamil NS (Part 2A). At least 18 subsequent patients will be enrolled and treated with the etripamil NS with the dose determined by the PK analysis and will undergo efficacy and safety/tolerability assessments (Part 2B).

The study will include the following visits: A Screening Visit, A Treatment Visit, , and A Follow-Up/End of Study Visit.

DETAILED DESCRIPTION:
NODE-202 is a Phase 2, multicenter, multinational, single-dose, open-label, 2-part, sequential design study of pediatric patients with an established diagnosis of PSVT presenting with a sustained, symptomatic episode of PSVT.

At least 60 evaluable patients administered etripamil NS are estimated as an adequate population to inform on the efficacy and safety of etripamil NS in pediatric patients (aged 6 to <18 years) with PSVT. Patients will be enrolled according to the following sequential design:

Part 1: At least 30 patients aged 12 to <18 years will be treated with 70 mg etripamil NS for a PSVT episode. Efficacy, safety, tolerability and PK (at least for 12 patients) will be assessed after administration of etripamil.

Part 1A: at least 12 patients will undergo efficacy, safety/tolerability, and PK assessments. The data safety monitoring committee (DSMC) will complete an interim assessment of safety, tolerability; if the Sponsor decides to increase the dose above 70 mg for the remaining 18 patients, the Pediatric Committee (PDCO) and the Food and Drug Administration (FDA) will complete an interim assessment of efficacy, safety, tolerability, and PK data before additional patients in this age group can be treated with etripamil at the same or a modified dose level.

Part 1B: at least 18 subsequent patients will be treated with etripamil NS with the dose determined based on Part 1A data analysis and will undergo efficacy and safety/tolerability assessments.

Part 2: Clinical assessments in at least 30 patients aged 6 to <12 years will only be undertaken if, after a comprehensive review of safety, tolerability, efficacy, and PK data collected in patients aged 12 to <18 years, confirms a positive benefit-risk ratio in that age group, sufficient to permit administration of etripamil NS in the younger age group. The initial dose for Part 2 will be selected based on appropriate body size-based modelling, as well as safety/tolerability, and efficacy data collected in Part 1.

Part 2A: at least 12 patients will undergo efficacy, safety/tolerability, and PK assessments. The DSMC will complete an interim assessment of safety, tolerability; the PDCO and FDA will complete an interim assessment of safety, tolerability, and PK data before additional patients in this age group can be treated with etripamil at the same or a modified dose level.

Part 2B: at least 18 subsequent patients will be enrolled and treated with etripamil NS with the dose determined based on Part 2A data analysis and will undergo efficacy and safety/tolerability assessments.

The study will include:

A Screening Visit during which the Investigator will verify that the patient currently meets the eligibility criteria of the NODE-202 study, will obtain the Informed Consent/Assent, will evaluate the patient's medical status and concomitant medications, will perform a 12-Lead ECG using provided study-specific equipment, will take blood and urine for clinical laboratory evaluations (local laboratory) and will assess the patient's eligibility according to the inclusion/exclusion criteria. Also, qualified patients will be instructed that as soon as they have identified symptoms they consider being consistent with PSVT, they must attend the Study Medical Facility assigned by their Investigator for a treatment visit.

A Treatment Visit during which patients will arrive at the Study Medical Facility with symptoms consistent with PSVT, and the following actions will be performed: confirmation of eligibility, evaluation of vital signs and initiation of a 12-lead Electrocardiogram (ECG) using the provided ECG equipment. If after ECG assessment diagnosis of PSVT is not confirmed, the patient must not be administered etripamil NS and will receive standard of care treatment based on the diagnosis. If ECG assessment confirms the presence of PSVT, a vagal maneuver (VM) will be performed by the patient or physician, based on the Investigator's judgement. If the VM is not successful in terminating the confirmed PSVT episode, etripamil NS will then be administered intranasally by study site personnel, under medical supervision and ECG monitoring for 1 hour.

A Follow-Up/End of Study Visit (1 to 5 days after an episode) during which any Adverse Events (AEs) and ECG will be recorded, and vital signs will be measured.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for study participation if they meet all of the following criteria at screening:

1. Male or female patients

   1. Part 1: patients 12 to <18 years of age
   2. Part 2: patients 6 to <12 years of age
2. Body mass index (BMI) between the 5th and the 85th percentiles interpreted relative sex and age
3. History of PSVT documented by ECG or other monitoring modality (e.g., Holter monitor, event recorder) showing SVT involving the Atrioventricular (AV) node (i.e., Atrioventricular nodal reentry tachycardia (AVNRT) or Atrioventricular reentrant tachycardia (AVRT)). If patient had a prior ablation for PSVT, patient must have documented evidence of PSVT post-ablation
4. Signed written informed consent/assent obtained
5. Per Investigator's decision, females of childbearing potential (defined as any woman or adolescent who has begun menstruation) must additionally satisfy the following criteria:

   1. Negative pregnancy test at screening
   2. Adequate contraception, unless total abstinence is used
6. Willing and able to comply with study procedures.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. History or presence of any of the following at the screening visit:

   1. Patients with a history of atrial arrhythmia that does not involve the AV node as part of the tachycardia circuit (e.g., atrial fibrillation, atrial flutter, atrial tachycardia) are not eligible
   2. Permanent junctional reciprocating tachycardia
   3. Ventricular pre-excitation (e.g., delta wave on ECG, Wolff Parkinson White syndrome)
   4. Second- or third-degree AV block
   5. Sick sinus syndrome or clinically significant bradycardia (<50 bpm or equivalent in this patient population) on the resting ECG
   6. Ventricular tachycardia
   7. Long QT syndrome
   8. Major structural heart disease (e.g., Ebstein's anomaly, corrected congenital heart disease) or symptoms of congestive heart failure (New York Heart Association class II to IV).
2. Evidence of impaired liver function (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST] >3 x upper limit of normal for age and gender) at the Screening Visit
3. Evidence of End-Stage Renal Disease as determined by an estimated glomerular filtration rate assessed at the Screening Visit of <15 mL/min/1.73m2, or requiring hemodialysis;
4. Treatment with any of the following that cannot or will not be discontinued during study participation:

   1. Any investigational drug within 60 days prior to study drug administration
   2. IV beta-adrenergic blocking drugs (e.g., propranolol, esmolol), calcium channel blocking drugs (e.g., verapamil, diltiazem) or amiodarone within 24 hours prior to study drug administration
   3. Oral amiodarone within 30 days prior to study drug administration
   4. Class I or III antiarrhythmic agents (e.g., flecainide, propafenone, sotalol) within five half-lives prior to study drug administration
   5. Any other drug that has a contraindication with verapamil
5. Known hypersensitivity to verapamil or to any of the excipients of the study drug
6. Any other significant co-morbid condition that may have a negative impact on the patient's participation in the study or likely to result in non-compliance
7. History of hyperthyroidism
8. Current pregnancy or breastfeeding

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy: The percentage of patients converting to sinus rhythm (SR) in the first 15 minutes after administration of etripamil NS. | 15 minutes after administration of etripamil NS
  A successful conversion is defined as conversion of PSVT to SR that is maintained for at least 30 seconds

SECONDARY OUTCOMES:
Efficacy: Time to termination of the PSVT episode and conversion to SR | 60 minutes after administration of etripamil NS
  Time measured from time of dosing to time of conversion of PSVT to SR that is maintained for at least 30 seconds
Efficacy: Percentage of patients requiring additional medical intervention treatment for the PSVT episode in the first 15 minutes after study drug administration. | 15 minutes after administration of etripamil NS
  Medical intervention is defined as an administered drug or procedure to treat PSVT
Safety: Frequency of AEs | Until 5 days after administration of etripamil NS
  Adverse Events (AEs) defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related
Safety: Local (administration site) tolerability | Until 5 days after administration of etripamil NS
  Local tolerability defined as frequency of adverse events related to nasal spray site administration
Safety: Post-dose changes in vital signs (Hearth rate (HR)) | Until 5 days after administration of etripamil NS
  HR changes as measured by increase/decrease in beats per minute
Safety: Post dose changes in vital sign (Blood Pressure (BP)) | Until 5 days after administration of etripamil NS
  BP changes (systolic blood pressure (SBP) and diastolic blood pressure (DBP)) as measured in increase/decrease in mmHg

OTHER OUTCOMES:
Pharmacokinetic analysis of etripamil: Maximum plasma concentration (Cmax) | Within 1 hour after administration of etripamil NS
  Maximum plasma concentration (Cmax) in ng/mL of etripamil assessed from PK analysis of plasma samples within 1 hour of dosing.
Pharmacokinetic analysis of etripamil: Area under the concentration-time curve from dosing (time 0) to time t (AUC0-t). | Within 1 hour after administration of etripamil NS
  Area under the concentration-time curve from dosing (time 0) to time t (AUC0-t) in min*ng/mL of etripamil assessed from PK analysis of plasma samples within 1 hour of dosing.
Pharmacokinetic analysis of etripamil: Area under the concentration-time curve from dosing (time 0) to time infinity (AUC0-inf). | Within 1 hour after administration of etripamil NS
  Area under the concentration-time curve from dosing (time 0) to time infinity (AUC0-inf) in min*ng/mL of etripamil assessed from PK analysis of plasma samples within 1 hour of dosing.
Pharmacokinetic analysis of etripamil: Elimination rate constant (Kel) | Within 1 hour after administration of etripamil NS
  Elimination rate constant (Kel) in 1/minutes of etripamil assessed from PK analysis of plasma samples within 1 hour of dosing.
Pharmacokinetic analysis of etripamil: Time to achieve maximum plasma concentration (tmax) | Within 1 hour after administration of etripamil NS
  Time to achieve maximum plasma concentration (tmax) in minutes of etripamil assessed from PK analysis of plasma samples within 1 hour of dosing.
Pharmacokinetic analysis of etripamil: Half-life (t1/2) | Within 1 hour after administration of etripamil NS
  Half-life (t1/2) in minutes of etripamil assessed from PK analysis of plasma samples within 1 hour of dosing.
Pharmacokinetic analysis of MSP-2030 (inactive metabolite): Maximum plasma concentration (Cmax) | Within 1 hour after administration of etripamil NS
  Maximum plasma concentration (Cmax) in ng/mL of MSP-2030 assessed from PK analysis of plasma samples within 1 hour of dosing.
Pharmacokinetic analysis of MSP-2030 (inactive metabolite): Area under the concentration-time curve from dosing (time 0) to time t (AUC0-t). | Within 1 hour after administration of etripamil NS
  Area under the concentration-time curve from dosing (time 0) to time t (AUC0-t) in min*ng/mL of MSP-2030 assessed from PK analysis of plasma samples within 1 hour of dosing.
Pharmacokinetic analysis of MSP-2030 (inactive metabolite): Area under the concentration-time curve from dosing (time 0) to time infinity (AUC0-inf). | Within 1 hour after administration of etripamil NS
  Area under the concentration-time curve from dosing (time 0) to time infinity (AUC0-inf) in min*ng/mL of MSP-2030 assessed from PK analysis of plasma samples within 1 hour of dosing.
Pharmacokinetic analysis of MSP-2030 (inactive metabolite): Elimination rate constant (Kel). | Within 1 hour after administration of etripamil NS
  Elimination rate constant (Kel) in 1/minutes of MSP-2030 assessed from PK analysis of plasma samples within 1 hour of dosing.
Pharmacokinetic analysis of MSP-2030 (inactive metabolite): Time to achieve maximum plasma concentration (tmax). | Within 1 hour after administration of etripamil NS
  Time to achieve maximum plasma concentration (tmax) in minutes of MSP-2030 assessed from PK analysis of plasma samples within 1 hour of dosing.
Pharmacokinetic analysis of MSP-2030 (inactive metabolite): Half-life (t1/2) | Within 1 hour after administration of etripamil NS
  Half-life (t1/2) in minutes of MSP-2030 assessed from PK analysis of plasma samples within 1 hour of dosing.

CONTACTS AND LOCATIONS:
Overall Officials: David Bharucha, MD, Study Director — Milestone Pharmaceuticals
Locations (10):
- United States (6):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Advocate Children's Hospital, Oak Lawn, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
- The University of British Columbia, Vancouver, Canada
- Universitätsmedizin Göttingen, Klinik für Pädiatrische Kardiologie, Intensivmedizin und Neonatologie, Göttingen, Germany
- Spain (2):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Infantil Universitario La Paz, Madrid